CLINICAL TRIAL: NCT03971981
Title: Xylitol Chewing-gums: Concentration in Saliva and Antibacterial Effect (In-vivo and In-vitro Study)
Brief Title: Xylitol Chewing-gums: Concentration in Saliva and Antibacterial Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Professor of Public Health Dentistry, Università degli Studi di Sassari
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SS-15884-GC
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Dental Caries; Periodontal Diseases
Keywords: Xylitol; Saliva; Bacteria; Dental Plaque; Antimicrobial effect; Chewing gum
MeSH Terms: conditions — Dental Caries; Periodontal Diseases; Dental Plaque

STUDY DESIGN:
Intervention Model Description: a double-blind cross-over in vivo study was performed to measure the salivary concentration of Xylitol released from the two chewing gums containing different amount of the polyol. The study had a cross-over design: the first half of the sample used the chewing-gum with Xylitol as the only sweeteners (64.5% of chewing-gum weight) and the other half use the chewing-gum with Xylitol among the sweeteners (22% of chewing-gum weight), after a 7-days wash-out period, the two sub-groups inverted the chewing gums. Subjects were instructed to consume the products as they normally would be consumed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100% Xylitol (Experimental): The study had a cross-over design: the first half of the sample used the chewing-gum with Xylitol as the only sweeteners (64.5% of chewing-gum weight) and the other half use the chewing-gum with Xylitol among the sweeteners (22% of chewing-gum weight), after a 7-days wash-out period, the two sub-groups inverted the chewing gums.
  Interventions: Dietary Supplement: 100% Xylitol Gum
- 22% Xylitol (Experimental): The study had a cross-over design: the first half of the sample used the chewing-gum with Xylitol as the only sweeteners (64.5% of chewing-gum weight) and the other half use the chewing-gum with Xylitol among the sweeteners (22% of chewing-gum weight), after a 7-days wash-out period, the two sub-groups inverted the chewing gums.
  Interventions: Dietary Supplement: 22% Xylitol Gum

INTERVENTIONS:
Dietary Supplement: 100% Xylitol Gum — Subjects were instructed to consume the gums as they normally would be consumed.
  Arms: 100% Xylitol
Dietary Supplement: 22% Xylitol Gum — Subjects were instructed to consume the gums as they normally would be consumed.
  Arms: 22% Xylitol

SUMMARY:
a double-blind cross-over in vivo study was performed to measure the salivary concentration of Xylitol released from the two chewing gums containing different amount of the polyol. The study had a cross-over design: the first half of the sample used the chewing-gum with Xylitol as the only sweeteners (64.5% of chewing-gum weight) and the other half use the chewing-gum with Xylitol among the sweeteners (22% of chewing-gum weight), after a 7-days wash-out period, the two sub-groups inverted the chewing gums. Subjects were instructed to consume the products as they normally would be consumed.

DETAILED DESCRIPTION:
x

ELIGIBILITY:
Inclusion Criteria:

* good general health,
* the absence of diseases that can alter the saliva secretion rate
* a stimulated saliva flow at least of 1 ml/min.

Exclusion Criteria:

-

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Change of Salivary concentration of Xylitol | 9 days
  Xylitol concentration using spectrophotometer analysis was determined in saliva before, at 0.30, 1.00, 2.00, 5.00, 10.00 minutes using the chewing-gum, and after the gum discarded at 15.00, 20.00 and 25.00 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Campus, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Department of Surgery, Microsurgery and Medicine Sciences University of Sassari, Sassari, Sardinia, Italy

IPD SHARING:
Plan to Share IPD: No